CLINICAL TRIAL: NCT05238259
Title: Kinesiotaping Versus Wrist Wheel on Upper Extremity Functions in Children With Hemiparetic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: Ministry of Health and Population, Egypt (Other Government)
Responsible Party: Principal Investigator, Mohamed Abd Elfatah Abd Elkarim Ibrahim, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KT versus Wrist wheel on Hemi
Record Dates: First submitted 2021-11-02; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Hemiplegic Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiotaping (Other): Kinesio tape is the name of an adhesive tape created by Kenzo Kase in Japan in 1973. Kinesiotaping is latex-free with 100% cotton fibers that has no pharmaceutical effect, designed to mimic the elasticity properties of the muscle, skin, and fascia. These properties make it resistant and wearable for a long period, in general, 3 to 5 days at a time; it is even water resistant.
  Interventions: Device: kinesiotaping
- wrist wheel (Other): Wrist wheel is a therapy aid that exercises muscles in the wrist, forearm and shoulder. It utilizes exercises known as pronation and supination moving from pronation to supination exercises is made easy because of the wheel. It allows the patient to easily roll wrist back and forth focusing on the wrist and arm
  Interventions: Device: wrist wheel

INTERVENTIONS:
Device: kinesiotaping — Kinesio tape is the name of an adhesive tape created by Kenzo Kase in Japan in 1973. Kinesiotaping is latex-free with 100% cotton fibers that has no pharmaceutical effect, designed to mimic the elasticity properties of the muscle, skin, and fascia. These properties make it resistant and wearable for a long period, in general, 3 to 5 days at a time; it is even water resistant.
  Arms: kinesiotaping
Device: wrist wheel — Wrist wheel is a therapy aid that exercises muscles in the wrist, forearm and shoulder. It utilizes exercises known as pronation and supination moving from pronation to supination exercises is made easy because of the wheel. It allows the pateint to easily roll wrist back and forth focusing on the wrist and arm
  Arms: wrist wheel

SUMMARY:
Investigate the effect of wrist wheel exercise on ROM of forearm supination and its reflection on upper extremity functions of children with HCP and Compare between effects of kinesiotaping and wrist wheel on ROM of forearm supination and its reflection on upper extremity functions of children with HCP

DETAILED DESCRIPTION:
Hemiparetic CP affects one side of the body, typically with marked involvement of the upper extremity, and is associated with reduced selective motor control and limited forearm supination . Hemiparetic child has a significant reduction of the effective use of the arm and hand in ADL (e.g. drinking, eating, accomplishing self-care, combing hair or dressing), and their participation at home, school, and later vocational roles .

Finding a therapeutic modality to improve ROM of forearm supination is an issue of concern in this study as a child uses varying degrees of supination throughout the day to complete simple activities. Some tasks only involve a person to use half of their supination ROM (e.g: clapping hands together) while other activities require a person to supinate through their full ROM (e.g: carrying a lunch tray). Hemiparetic child has limited supination movement, therefore this study will be conducted to investigate and compare between the therapeutic outcomes of kinesiotaping and wrist wheel on ROM of forearm supination which is important for upper extremity functions of the children with HCP.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from six to eight years.
* Diagnosed as HCP.
* Children with mild upper limb spasticity in all upper limb muscles (grades 1 to 1+) according to modified Ashworth scale.
* Children had impaired hand functions level II and III according to Manual Ability Classification System.
* They had the ability to follow simple verbal commands regarding assessment and treatment

Exclusion Criteria:

* Sever visual or auditory problems
* Children with severe sensory at the affected upper limb.
* Recent orthopedic surgical interference in the affected upper limb in the last six months before the study (Tenotomy or muscle transfer in the affected upper limb)
* Recent botulinum toxin injection of the affected upper extremity muscles in the last six months before the study.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Digital Goniometer used to measure range of motion of forearm supination in Children with Hemiparetic Cerebral Palsy. | baseline
  48 children from both genders participated in this study.They assessed by Digital Goniometer to measure range of motion of forearm supination in Children with Hemiparetic Cerebral Palsy.They selected by Modified Ashworth Scale to rate muscle spasticity that all subjects selected in this study are graded 1 to 1+ for affected upper limb muscles and Manual Ability Classification System that all subjects selected in this study level II and III .
Shriners Hospital Upper Extremity Evaluation (SHUEE) used to evaluate the spontaneous use of the involved extremity and evaluate the segmental alignment of the extremity while performing tasks on demand in Children with Hemiparetic Cerebral Palsy. | baseline
  48 children from both genders participated in this study.They assessed by Shriners Hospital Upper Extremity Evaluation (SHUEE) to evaluate upper extremity functions in Children with Hemiparetic Cerebral Palsy.They selected by Modified Ashworth Scale to rate muscle spasticity that all subjects selected in this study are graded 1 to 1+ for affected upper limb muscles and Manual Ability Classification System that all subjects selected in this study level II and III .

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Abd Elfatah abd El karim Ibrahim, Cairo, Egypt

REFERENCES:
- [Background] Shamsoddini A, Rasti Z, Kalantari M, Hollisaz MT, Sobhani V, Dalvand H, Bakhshandeh-Bali MK. The impact of Kinesio taping technique on children with cerebral palsy. Iran J Neurol. 2016 Oct 7;15(4):219-227. PMID 28435631
- [Background] Allah RASTIl Z, Shamsoddini A, Dalvand H, Labaf S. The Effect of Kinesio Taping on Handgrip and Active Range of Motion of Hand in Children with Cerebral Palsy. Iran J Child Neurol. 2017 Fall;11(4):43-51. PMID 29201123